CLINICAL TRIAL: NCT01142414
Title: Randomized Phase III Trial on Postoperative Chemoradiation in Combination With Anti EGFR-Antibody Versus Postoperative Chemoradiation in Head and Neck Squamous Cell Carcinomas (HNSCC) With High Risk of Locoregional Recurrence
Brief Title: Chemotherapy and Radiation Therapy With or Without Panitumumab in Treating Patients Who Have Undergone Surgery for Advanced Hypopharyngeal Cancer, Oropharyngeal Cancer, Laryngeal Cancer, or Oral Cavity Cancer at High Risk of Recurrence
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-22071-24071; EORTC-22071; EORTC-22071-24071; EU-21038; EUDRACT-2008-006180-36; AMGEN-EORTC-22071
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Panitumumab; Cisplatin; Fluorouracil; Chemotherapy, Adjuvant; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Biological: panitumumab
Drug: cisplatin
Drug: fluorouracil
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: quality-of-life assessment
Radiation: 3-dimensional conformal radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether chemotherapy given together with radiation therapy is more effective with or without panitumumab in treating patients with advanced cancer of the hypopharynx, oropharynx, larynx, or oral cavity.

PURPOSE: This randomized phase III trial is studying chemotherapy given together with radiation therapy to see how well it works compared with chemotherapy and radiation therapy given together with panitumumab in treating patients who have undergone surgery for advanced hypopharyngeal cancer, oropharyngeal cancer, laryngeal cancer, or oral cavity cancer at high risk of recurrence.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the addition of concurrently administered panitumumab to standard adjuvant chemoradiation, with 1 of 2 cisplatin-based regimens, significantly prolongs disease-free survival of patients with macroscopically completely resected, advanced squamous cell carcinoma of the hypopharynx, oropharynx, larynx, or oral cavity at high risk of recurrence.

Secondary

* To determine if the pre-surgery dose of panitumumab will alter the RNA expression of several genes and that these changes will provide additional prognostic information that can be used in future patient management. (Exploratory)
* Measure the differences in RNA expression by RNA microarray and the results analyzed to create a gene expression classifier that will be checked for outcome prediction by association with disease free survival and down regulation of the glucose metabolism as measured by FDG-PET. (Exploratory)
* To create a European biobank of biological samples which can be used for future research projects in this disease. (Exploratory)
* To predict radiation-induced normal tissue toxicity based on in vitro lymphocyte apoptosis test and SNPs analysis. (Exploratory)
* To assess the impact of radiation-induced side effects (swallowing dysfunction and xerostomia) on patient's quality of life.

OUTLINE: This is a multicenter study. Patients are stratified by treatment center, radiotherapy technique (3D-CRT vs IMRT), chemotherapy regimen (European Organization for Research and Treatment of Cancer [EORTC]) vs Arbeitsgemeinschaft Radiology Oncology [ARO] schedule), tumor location (larynx vs oropharynx vs hypopharynx vs oral cavity), pN-stage (pN0-2 vs pN3), pT-stage (pT1-2 vs pT3-4), margin/extracapsular extension (ECE) status (ECE+ and margin < 5 mm vs ECE- and margin < 5 mm vs ECE+ and margin > 5 mm), biological pre-study participation (yes vs no), p16 status (positive vs negative vs indeterminable). Patients are randomized to 1 of 2 treatment arms.

* Arm I (chemoradiotherapy): Within 4-8 weeks of surgery, patients undergo 3D-conformal or intensity-modulated radiotherapy once daily 5 days a week in weeks 1-7. Patients also receive concurrent chemotherapy comprising either cisplatin IV over 1-2 hours on days 1, 22, and 43 (EORTC schedule) OR cisplatin IV over 1-2 hours and fluorouracil IV over 24 hours on days 1-5 and 29-33 (ARO schedule), in the absence of disease progression or unacceptable toxicity.
* Arm II (chemoradiotherapy plus panitumumab): Within 4-8 weeks of surgery, patients undergo 3D-conformal or intensity-modulated radiotherapy and receive concurrent chemotherapy (EORTC schedule or ARO schedule) as in arm I. Patients also receive panitumumab IV over 1 hour on days 1, 8, 15, 22, 29, 36, and 43.

Blood samples are collected periodically for biomarker correlative studies and translational research. Patients complete quality-of-life EORTC questionnaires QLQ-C30, QLQ-HN35, and PSS-HN periodically.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary squamous cell carcinoma of the hypopharynx, oropharynx, larynx, or oral cavity

  * Stage pT1-2 pN+ or pT3-4 any pN (stage III-IVB) disease
  * No distant metastases
  * No recurrent disease
* Resectable disease

  * Has undergone surgical resection of carcinoma

    * p16 immunohistochemistry assay performed on tissue sections taken during the surgical procedure
    * No laser surgery
* Potentially at high-risk of locoregional recurrence, defined as fulfilling ≥ 1 of the following criteria:

  * Close surgical margins (i.e., margins 1 mm to < 5 mm)
  * R1-resection (< 1 mm) (R2 resection is considered as not eligible)
  * Extracapsular nodal extension
* No nasopharynx, nasal cavity, or paranasal sinuses carcinomas

PATIENT CHARACTERISTICS:

* WHO or ECOG performance status 0-1
* Absolute neutrophils ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 10.0 g/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST< 3 times ULN
* Alkaline phosphatase < 3 times ULN
* Calculated creatinine clearance ≥ 60 mL/min
* Calcium ≤ 11.5 mg/dL or 2.9 mmol/L
* Magnesium ≥ 1.2 mg/dL or 0.5 mmol/L
* Fertile patients must use effective contraception methods during the study and for 6 months after the last treatment dose
* Not pregnant or nursing
* No known allergic or hypersensitivity reaction to any of the components of the study treatment
* No other concurrent serious illnesses or medical conditions, including any of the following:

  * History or evidence of interstitial pneumonitis or pulmonary fibrosis
  * Unstable cardiac disease despite treatment
  * NYHA class III-IV congestive heart failure
  * Clinically significant abnormal ECG or LVEF below the institutional lower limit of normal
  * Known HIV infection or other conditions of persistent immunodeficiency
  * Significant neurologic or psychiatric disorders
  * Active uncontrolled infection
  * Active disseminated intravascular coagulation
  * Symptomatic peripheral neuropathy (CTCAE 4.0 "peripheral sensory neuropathy and paresthesia") ≥ grade 2 or ototoxicity (CTCAE 4.0 "hearing impaired") ≥ grade 2, unless due to trauma or mechanical impairment due to tumor mass
  * Other serious underlying medical conditions that could impair the ability of the patient to participate in the study
* No other malignancy within the past 5 years other than basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix

  * Patients who are disease-free for > 5 years allowed
* No known drug abuse
* No psychological, familial, sociological (e.g., severe alcohol addiction expected to hamper protocol compliance), or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for carcinoma of the head and neck
* No prior radiotherapy to the head and neck region
* No prior exposure to EGFR pathway-targeting therapy
* No participation in another interventional clinical trial within the past 30 days
* No concurrent granulocyte colony-stimulating factor (G-CSF) or erythropoietin
* No other concurrent investigational drugs and/or anticancer treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival
Loco-regional control
Cumulative incidence of and time to distant metastases
Cumulative incidence of and time to second cancers (all sites)
Incidence of acute and late toxicity (CTCAE version 4.0)
Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Budach, MD, Study Chair — Heinrich-Heine University, Duesseldorf; Hans Langendijk, Study Chair — University Medical Center Groningen; Carla Van Herpen, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen

REFERENCES:
- [Result] Liberatoscioli C, Langendijk JA, Van Herpen C, et al.: EORTC 22071-24071: randomized, phase III trial of EGFR-antibody combined with adjuvant chemoradiation for patients with head and neck squamous cell carcinoma (HNSCC) at high risk of recurrence. [Abstract] J Clin Oncol 29 (Suppl 15): A-TPS197, 2011.